CLINICAL TRIAL: NCT02480218
Title: Cognitive Sequelae of Adjuvant Endocrine Therapy for the Treatment of Breast Cancer in Older Women
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 130-2015
Record Dates: First submitted 2015-06-11; First posted 2015-06-24 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
Keywords: cognition; tamoxifen; aromatase inhibitors
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tamoxifen: Chemotherapy-naïve women 65 and older with a first diagnosis of early stage HR+ BC, post surgical resection prescribed tamoxifen.
  Interventions: Other: Neuropsychological test battery
- Aromatase Inhibitors: Chemotherapy-naïve women 65 and older with a first diagnosis of early stage HR+ BC, post surgical resection prescribed aromatase inhibitors.
  Interventions: Other: Neuropsychological test battery

INTERVENTIONS:
Other: Neuropsychological test battery — Participants will have been prescribed their endocrine therapy for the treatment of breast cancer prior to enrollment. Neuropsychological test batteries will be administered at baseline and at one-year follow-up to assess changes in cognition.

SUMMARY:
Breast cancer is the most frequently diagnosed cancer in women with the majority receiving an endocrine therapy (ET) in the adjuvant setting. ETs dramatically reduce recurrence and improve survival but given the aging population and increased survivorship, there are growing concerns regarding the cognitive effects of ETs since estrogen is neuroprotective. A critical unanswered question is whether there are differences in cognitive decline between the two classes of ETs, selective estrogen receptor modulators (SERMs - tamoxifen) and aromatase inhibitors (letrozole and anastrozole), in older women at greater risk of hormone receptor breast cancer and cognitive decline. Before a large multicentre observational study can be undertaken the investigators are proposing a feasibility study to establish metrics on participation, retention and adherence rates and parameter estimates to inform sample size calculation required to detect cognitive differences between the two ET classes. A convenience sample of chemotherapy-naïve patients, aged 65 and older, with early stage disease, 25 on a SERM and 50 on an aromatase inhibitor, will be assessed cognitively at baseline and after one year.

DETAILED DESCRIPTION:
The convenience sample will consist of chemotherapy-naïve women 65 and older with a first diagnosis of early stage HR+ BC, post surgical resection, who are prescribed either TAM (n=25) or an AI, anastrozole or letrozole (n=50). Based on a survey of medical oncologist prescribing practices at Sunnybrook, the investigators will be able to obtain sufficient numbers for the convenience sample from the pool of 220 older women with BC referred annually to medical and radiation oncology at the Louise Temerty Breast Cancer Clinic and the Odette Cancer Centre . The investigators will recruit consecutively seen eligible patients before radiotherapy. Experienced clinical trial staff will identify eligible patients from the clinic list of each medical and radiation oncologist, who will then introduce the study during the visit. The Research Coordinator (RC) will meet with interested patients for consent to conduct the screening assessment for signs of cognitive impairment using the Memory Impairment Screen (MIS), a sensitive and reliable tool. The MIS will take no more than 5 minutes and will be conducted in a private room at either the Louise Temerty Breast Cancer Centre or the Odette Cancer Centre depending on the location of the patient's appointment. The RC will then obtain consent from all those who pass the MIS to participate in the study and arrange for testing. The RC will administer the assessment battery at a time convenient to the patient, before radiotherapy. Drug adherence rates will be obtained using monthly telephone self-reports. After 1 year, participants will undergo the same testing protocol as at baseline using alternate forms where possible. The RC will document how many continue to meet study criteria including changes in health status, medications, etc. The investigators do not expect any major selection biases between our groups. While exclusion of women co-administered chemotherapy due to its confounding effects on cognition may bias the sample by including more women with co-morbidities, this potential bias should be reduced by our exclusion of previous cancers, life expectancy <2 years, and central nervous system (CNS) disorders. To determine bias in attrition of women at year 1 due to cognitive impairment, the investigators will contact all participants and caregivers who do not return to determine the reason.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female, age 65 and older
* No more than 14 weeks post surgical resection for early stage histologically confirmed hormone receptor positive (HR+) breast cancer (BC) (i.e., Tumour size 1-2, Node status 0-1, Metastasis 0). HR+ BC defined as >1% positive cell staining
* Prescribed either tamoxifen, letrozole, or anastrozole
* Fluent in written and spoken English; >grade 5 education; can read large print (with or without correction); can hear normal conversation (with or without a hearing aid)
* Capacity to provide informed consent

Exclusion Criteria:

* Initiated adjuvant ET more than one week before baseline assessment
* Chemotherapy (neoadjuvant or adjuvant)
* More than one treatment of radiotherapy before baseline assessment
* Hormone replacement therapy use 4 weeks prior to baseline assessment
* Previous breast cancer or metastatic disease or other malignancy, other than any cancers treated for cure >5 years ago and not having recurred except non-melanoma skin cancers; previous chemotherapy; previous use of selective estrogen receptor modulators (SERM) or aromatase inhibitor (AI); distant metastases
* History of or active known CNS disease (e.g. known diagnosis of stroke, Parkinson's), medical condition impairing cognitive function, including active treatment with medication known to affect cognition, or signs of cognitive impairment on the Memory Impairment Screen
* History or active known diagnosis of major psychiatric disorder in the last 10 years including bipolar disease, schizophrenia, major depression or self-reported hospitalization for psychiatric illness, alcoholism, or history of alcohol or drug abuse
* Life expectancy less than two years, acutely ill or delirious

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: chemotherapy-naïve women 65 and older with a first diagnosis of early stage HR+ BC, post surgical resection, who are prescribed either tamoxifen, anastrozole or letrozole.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who experience cognitive impairment after 1 year of treatment | 1 year
  Cognitive impairment will be defined as scoring at or below -1.5 standard deviations from the normative mean on two or more tests, or as scoring at or below -2.0 standard deviations on a single test.

CONTACTS AND LOCATIONS:
Overall Officials: Mary C. Tierney, PhD, Principal Investigator — Sunnybrook Health Sciences Centre; Kathleen Pritchard, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada